CLINICAL TRIAL: NCT05247840
Title: INvesTigation the Abnormality of Detrusor ConTractility by Uroflowmetry in Diabetic Children (INTACT Trial) - a Prospective, Cross-sectional, Observational, Controlled Study
Brief Title: INTACT Trial - an Observational Study to Assess Neuropathy in Diabetic Children
Acronym: INTACT
Status: Not yet recruiting | Type: Observational
Sponsor: Heim Pal Children's Hospital (Other)
Responsible Party: Principal Investigator, László Szabó MD, PhD, med habil., Prof. Dr. László Szabó M.D., PhD., DSc., Dr., Habil. pediatric nephrologist, urodynamic specialist, Heim Pal Children's Hospital
Other Study IDs: KUT-37/2021
Record Dates: First submitted 2022-01-18; First posted 2022-02-21 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; uroflowmetry; neuropathy; paediatric; children
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic children: Children aged 5-18 years (boys, girls) with type 1, type 2 and monogenic diabetes mellitus who are treated at the Endocrinology Department and Outpatient Clinic of Heim Pál National Pediatric Institute (HOGYI, Budapest, Hungary) will be enrolled. Definition of diabetes is based on the American Diabetes Association (ADA) criteria. All patients who meet the inclusion criteria will be informed of the possibility of taking part in the INTACT Trial.
  Interventions: Diagnostic Test: uroflowmetry; Diagnostic Test: Cardiovascular autonomic dysfunction test proposed by Ewing et al.; Diagnostic Test: peripheral nerve conduction test
- healthy children: Healthy children aged 5-18 years (boys, girls) without any acute or chronical disease will be will enrolled and the same tests will be performed on them as in diabetic children. Children with voided volume <20 mL, postvoid residual volume >15%, and signs of an overstretched bladder [voided volume more than: 30 x age (years) + 30 mL] will be excluded.
  Interventions: Diagnostic Test: uroflowmetry; Diagnostic Test: Cardiovascular autonomic dysfunction test proposed by Ewing et al.; Diagnostic Test: peripheral nerve conduction test

INTERVENTIONS:
Diagnostic Test: uroflowmetry — Uroflowmetry will be performed using a uroflow-cystometer (UroDoc Frytech) which determines Qmax, Qave and TQmax. Voided volume (in mL), voiding time (in sec), average and maximum urinary flow rate (Qave and Qmax in mL/sec), and time to maximum urinary flow (TQmax in sec) will be measured; urine flow acceleration (Qacc in mL/sec2) will be calculated. Qmax and Qave are defined according to the International Children's Continence Society. Voided volume will be measured by the uroflow-cystometer device; boys void in a standing, girls in a sitting position. Postvoid bladder diameter (mm) will be measured by ultrasonography and converted to bladder residual volume (mL). The device will be calibrated according to the prescribed instructions for use by a skilled technician. The examinations will take approximately 10 minutes.
  Other Names: non-invasive urodynamic test
Diagnostic Test: Cardiovascular autonomic dysfunction test proposed by Ewing et al. — CAD will be assessed by five reproducible and standardized cardiovascular reflex tests described by Ewing et al. Three of the five tests assess parasympathetic function: heart rate response to deep breathing, to standing, and the Valsalva maneuver. Two tests evaluate sympathetic function which are blood pressure responses from lying to standing and at sustained handgrip. Each of these five tests is assigned a score of 0 for normal, 0.5 for borderline, and 1 for abnormal results. The sum of these 5 scores - which is the Ewing score - is used to assess severity of CAD. Patients having Ewing score ≥ 2 form the CAD + group, and patients who have less than 2 form the CAD - group.
Diagnostic Test: peripheral nerve conduction test — Peripheral neuropathy will be evaluated by nerve conduction test. The device measures motor conduction in the lower extremities. It operates at two dedicated frequencies in order to perform a thick myelin sheath cordless fibre (5Hz) and thin myelinated nerve fibre (2000Hz) examination. The device will be calibrated according to the prescribed instructions for use by a skilled technician.

SUMMARY:
It is a prospective, cross-sectional, observational, controlled, single centre clinical study. Diabetic patients fulfilling the inclusion criteria and healthy controls will have uroflowmetry examination, cardiovascular autonomic dysfunction tests (heart rate response to deep breathing, to Valsalva maneuver, blood pressure and heart rate response to standing up, and to sustained handgrip), and peripheral nerve conduction test. The primary endpoint is the diagnostic accuracy (sensitivity, specificity, negative and positive predictive values) of the tests. The secondary endpoints are: differences in metabolic status (weight, height, body surface, BMI, laboratory parameters, body composition), fluid turnover, and clinical symptoms of diabetic patients comparing to healthy children.

DETAILED DESCRIPTION:
The autonomic nervous system function is examined by the reproducible and standardized cardiovascular reflex tests described by Ewing et al.. During the examination, electrocardiogram and blood pressure values are recorded continuously. Heart rate response to deep inspiration is executed to investigate the parasympathetic nervous system. Peripheral neuropathy is evaluated by nerve conduction test.

The trial will start with a pilot period, when the first 50 diabetic and 50 healthy children will be assessed. This will be followed by a short evaluation period, during which the principal investigators and the study team could make adjustments in the study protocol to ensure feasibility.

ELIGIBILITY:
Inclusion Criteria:

* 5-18 years (boys, girls) with type 1, type 2 and monogenic DM

Exclusion Criteria:

1. Acute febrile condition (≥38 °C core temperature) in the past seven days
2. Acute or chronical urinary tract or kidney disease: renal insufficiency (GFR ≤ 60 mL/min per 1.73 m2, urinary tract infection
3. Urological disease: bladder cancer, urolithiasis, urethral stricture, posterior urethral valve, meatal stenosis, previous genitourinary surgery, conditions causing urinary outflow problems (phimosis, hypospadias, vesicoureteral reflux)
4. Cystic fibrosis-related diabetes (CFRD)
5. Neurological disorders (multiple sclerosis, transient ischaemic attack, transverse myelitis, myelocele, meningomyelocele, previous spinal cord operation, or operation which might injure the sacral nerve plexus)
6. Medicines taken which can cause neuropathy:

   1. Cytostatic agents: cyclophosphamide, platinum-based antineoplastic agents, vinca alkaloids, epothilones, taxanes, proteasome inhibitors, immunomodulatory drugs
   2. Immunosuppressive agents: TNF-alfa inhibitors (adalimumab, infliximab, etanercept), interferon
   3. Cardiovascular medicines: statins, digoxin, amiodaron
   4. Antimicrobial agents: nitrofurantoin, linezolid, voriconazole, itraconazole, antituberculotics, metronidazole, fluoroquinolone
   5. Anti-ulcerative agent: cimetidin
   6. Neuropsychological agents: levodopa, fenitoin
7. Psychiatric disorders that prevents participation / collaboration in the study
8. Constipation (defined according to the Rome IV criteria)
9. Voided volume <20 mL
10. Patients who are pregnant, or gave birth in the last 12 months
11. Lack of consent of the patient or legal representative; the patient or legal representative withdraws his or her voluntary consent during the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Diabetic patients who are treated at the Endocrinology Department and Outpatient Clinic of Heim Pál National Pediatric Institute (HOGYI, Budapest, Hungary) will be enrolled.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of uroflowmetry test 1.1 | baseline
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of uroflowmetry test 1.2 | change from baseline at 12 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of uroflowmetry test 1.3 | change from baseline at 24 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of uroflowmetry test 1.4 | change from baseline at 36 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of uroflowmetry test 1.5 | change from baseline at 48 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of uroflowmetry test 1.6 | change from baseline at 60 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of cardiovascular autonomic dysfunction test 2.1 | baseline
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of cardiovascular autonomic dysfunction test 2.2 | change from baseline at 12 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of cardiovascular autonomic dysfunction test 2.3 | change from baseline at 24 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of cardiovascular autonomic dysfunction test 2.4 | change from baseline at 36 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of cardiovascular autonomic dysfunction test 2.5 | change from baseline at 48 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of cardiovascular autonomic dysfunction test 2.6 | change from baseline at 60 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of peripheral nerve conduction test 3.1 | baseline
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of peripheral nerve conduction test 3.2 | change from baseline at 12 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of peripheral nerve conduction test 3.3 | change from baseline at 24 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of peripheral nerve conduction test 3.4 | change from baseline at 36 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of peripheral nerve conduction test 3.5 | change from baseline at 48 months
  sensitivity, specificity, positive predictive value, negative predictive value
diagnostic accuracy of peripheral nerve conduction test 3.6 | change from baseline at 60 months
  sensitivity, specificity, positive predictive value, negative predictive value

SECONDARY OUTCOMES:
metabolic status 1.1 | baseline
  weight (kg)
metabolic status 1.2 | change from baseline at 12 months
  weight (kg)
metabolic status 1.3 | change from baseline at 24 months
  weight (kg)
metabolic status 1.4 | change from baseline at 36 months
  weight (kg)
metabolic status 1.5 | change from baseline at 48 months
  weight (kg)
metabolic status 1.6 | change from baseline at 60 months
  weight (kg)
metabolic status 2.1 | baseline
  height (cm)
metabolic status 2.2 | change from baseline at 12 months
  height (cm)
metabolic status 2.3 | change from baseline at 24 months
  height (cm)
metabolic status 2.4 | change from baseline at 36 months
  height (cm)
metabolic status 2.5 | change from baseline at 48 months
  height (cm)
metabolic status 2.6 | change from baseline at 60 months
  height (cm)
metabolic status 3.1 | baseline
  body surface (m2 calculated by the Mosteller formula)
metabolic status 3.2 | change from baseline at 12 months
  body surface (m2 calculated by the Mosteller formula)
metabolic status 3.3 | change from baseline at 24 months
  body surface (m2 calculated by the Mosteller formula)
metabolic status 3.4 | change from baseline at 36 months
  body surface (m2 calculated by the Mosteller formula)
metabolic status 3.5 | change from baseline at 48 months
  body surface (m2 calculated by the Mosteller formula)
metabolic status 3.6 | change from baseline at 60 months
  body surface (m2 calculated by the Mosteller formula)
metabolic status 4.1 | baseline
  BMI (kg/m2)
metabolic status 4.2 | change from baseline at 12 months
  BMI (kg/m2)
metabolic status 4.3 | change from baseline at 24 months
  BMI (kg/m2)
metabolic status 4.4 | change from baseline at 36 months
  BMI (kg/m2)
metabolic status 4.5 | change from baseline at 48 months
  BMI (kg/m2)
metabolic status 4.6 | change from baseline at 60 months
  BMI (kg/m2)
metabolic status 5.1 | baseline
  body composition evaluated by the Inbody device
metabolic status 5.2 | change from baseline at 12 months
  body composition evaluated by the Inbody device
metabolic status 5.3 | change from baseline at 24 months
  body composition evaluated by the Inbody device
metabolic status 5.4 | change from baseline at 36 months
  body composition evaluated by the Inbody device
metabolic status 5.5 | change from baseline at 48 months
  body composition evaluated by the Inbody device
metabolic status 5.6 | change from baseline at 60 months
  body composition evaluated by the Inbody device
metabolic status 6.1 | baseline
  laboratory parameters (CRP, ESR, full blood count, Hemoglobin, hematocrit, thrombocyte, glucose, C-peptide, HbA1c, triglyceride, cholesterol, uric acid, creatinine, carbamide, AST, ALT, GGT, LDH, ALP, Na, K, P, Ca, albumin, serum total protein, lipase, amylase, urine rapid test)
metabolic status 6.2 | change from baseline at 12 months
  laboratory parameters (CRP, ESR, full blood count, Hemoglobin, hematocrit, thrombocyte, glucose, C-peptide, HbA1c, triglyceride, cholesterol, uric acid, creatinine, carbamide, AST, ALT, GGT, LDH, ALP, Na, K, P, Ca, albumin, serum total protein, lipase, amylase, urine rapid test)
metabolic status 6.3 | change from baseline at 24 months
  laboratory parameters (CRP, ESR, full blood count, Hemoglobin, hematocrit, thrombocyte, glucose, C-peptide, HbA1c, triglyceride, cholesterol, uric acid, creatinine, carbamide, AST, ALT, GGT, LDH, ALP, Na, K, P, Ca, albumin, serum total protein, lipase, amylase, urine rapid test)
metabolic status 6.4 | change from baseline at 36 months
  laboratory parameters (CRP, ESR, full blood count, Hemoglobin, hematocrit, thrombocyte, glucose, C-peptide, HbA1c, triglyceride, cholesterol, uric acid, creatinine, carbamide, AST, ALT, GGT, LDH, ALP, Na, K, P, Ca, albumin, serum total protein, lipase, amylase, urine rapid test)
metabolic status 6.5 | change from baseline at 48 months
  laboratory parameters (CRP, ESR, full blood count, Hemoglobin, hematocrit, thrombocyte, glucose, C-peptide, HbA1c, triglyceride, cholesterol, uric acid, creatinine, carbamide, AST, ALT, GGT, LDH, ALP, Na, K, P, Ca, albumin, serum total protein, lipase, amylase, urine rapid test)
metabolic status 6.6 | change from baseline at 60 months
  laboratory parameters (CRP, ESR, full blood count, Hemoglobin, hematocrit, thrombocyte, glucose, C-peptide, HbA1c, triglyceride, cholesterol, uric acid, creatinine, carbamide, AST, ALT, GGT, LDH, ALP, Na, K, P, Ca, albumin, serum total protein, lipase, amylase, urine rapid test)
metabolic status 7.1 | baseline
  fluid turnover in 24 hours (mL)
metabolic status 7.2 | change from baseline at 12 months
  fluid turnover in 24 hours (mL)
metabolic status 7.3 | change from baseline at 24 months
  fluid turnover in 24 hours (mL)
metabolic status 7.4 | change from baseline at 36 months
  fluid turnover in 24 hours (mL)
metabolic status 7.5 | change from baseline at 48 months
  fluid turnover in 24 hours (mL)
metabolic status 7.6 | change from baseline at 60 months
  fluid turnover in 24 hours (mL)
clinical symptoms of diabetic patients will be measured and compared to healthy children. 8.1 | baseline
  clinical symptoms (Urgent urination, Daily urine incontinence, Urination during night time, Nocturia, Frequency of bowel movement, Consistency of the stool)
clinical symptoms of diabetic patients will be measured and compared to healthy children. 8.2 | change from baseline at 12 months
  clinical symptoms (Urgent urination, Daily urine incontinence, Urination during night time, Nocturia, Frequency of bowel movement, Consistency of the stool)
clinical symptoms of diabetic patients will be measured and compared to healthy children. 8.3 | change from baseline at 24 months
  clinical symptoms (Urgent urination, Daily urine incontinence, Urination during night time, Nocturia, Frequency of bowel movement, Consistency of the stool)
clinical symptoms of diabetic patients will be measured and compared to healthy children. 8.4 | change from baseline at 36 months
  clinical symptoms (Urgent urination, Daily urine incontinence, Urination during night time, Nocturia, Frequency of bowel movement, Consistency of the stool)
clinical symptoms of diabetic patients will be measured and compared to healthy children. 8.5 | change from baseline at 48 months
  clinical symptoms (Urgent urination, Daily urine incontinence, Urination during night time, Nocturia, Frequency of bowel movement, Consistency of the stool)
clinical symptoms of diabetic patients will be measured and compared to healthy children. 8.6 | change from baseline at 60 months
  clinical symptoms (Urgent urination, Daily urine incontinence, Urination during night time, Nocturia, Frequency of bowel movement, Consistency of the stool)

CONTACTS AND LOCATIONS:
Locations (1):
- Heim Pal National Pediatric Institute, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petropoulos IN, Ponirakis G, Khan A, Almuhannadi H, Gad H, Malik RA. Diagnosing Diabetic Neuropathy: Something Old, Something New. Diabetes Metab J. 2018 Aug;42(4):255-269. doi: 10.4093/dmj.2018.0056. PMID 30136449
- [Background] Yuan Z, Tang Z, He C, Tang W. Diabetic cystopathy: A review. J Diabetes. 2015 Jul;7(4):442-7. doi: 10.1111/1753-0407.12272. Epub 2015 Mar 24. PMID 25619174
- [Background] Arrellano-Valdez F, Urrutia-Osorio M, Arroyo C, Soto-Vega E. A comprehensive review of urologic complications in patients with diabetes. Springerplus. 2014 Sep 23;3:549. doi: 10.1186/2193-1801-3-549. eCollection 2014. PMID 25332855
- [Background] Fayyad AM, Hill SR, Jones G. Prevalence and risk factors for bothersome lower urinary tract symptoms in women with diabetes mellitus from hospital-based diabetes clinic. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Nov;20(11):1339-44. doi: 10.1007/s00192-009-0949-z. Epub 2009 Jul 15. PMID 19603127
- [Background] Kaplan SA, Te AE, Blaivas JG. Urodynamic findings in patients with diabetic cystopathy. J Urol. 1995 Feb;153(2):342-4. doi: 10.1097/00005392-199502000-00013. PMID 7815578
- [Background] Agashe S, Petak S. Cardiac Autonomic Neuropathy in Diabetes Mellitus. Methodist Debakey Cardiovasc J. 2018 Oct-Dec;14(4):251-256. doi: 10.14797/mdcj-14-4-251. PMID 30788010
- [Background] Ewing DJ, Clarke BF. Autonomic neuropathy: its diagnosis and prognosis. Clin Endocrinol Metab. 1986 Nov;15(4):855-88. doi: 10.1016/s0300-595x(86)80078-0. PMID 3536203
- [Background] Barkai L, Szabo L. Urinary bladder dysfunction in diabetic children with and without subclinical cardiovascular autonomic neuropathy. Eur J Pediatr. 1993 Mar;152(3):190-2. doi: 10.1007/BF01956141. PMID 8444242
- [Background] Szabo L, Barkai L, Lombay B. Urinary flow disturbance as an early sign of autonomic neuropathy in diabetic children and adolescents. Neurourol Urodyn. 2007;26(2):218-21. doi: 10.1002/nau.20349. PMID 17078072
- [Background] Zajaczkowska R, Kocot-Kepska M, Leppert W, Wrzosek A, Mika J, Wordliczek J. Mechanisms of Chemotherapy-Induced Peripheral Neuropathy. Int J Mol Sci. 2019 Mar 22;20(6):1451. doi: 10.3390/ijms20061451. PMID 30909387
- [Background] Jones MR, Urits I, Wolf J, Corrigan D, Colburn L, Peterson E, Williamson A, Viswanath O. Drug-Induced Peripheral Neuropathy: A Narrative Review. Curr Clin Pharmacol. 2020;15(1):38-48. doi: 10.2174/1574884714666190121154813. PMID 30666914
- [Background] Ewing DJ, Martyn CN, Young RJ, Clarke BF. The value of cardiovascular autonomic function tests: 10 years experience in diabetes. Diabetes Care. 1985 Sep-Oct;8(5):491-8. doi: 10.2337/diacare.8.5.491. PMID 4053936
- [Background] Spallone V, Bellavere F, Scionti L, Maule S, Quadri R, Bax G, Melga P, Viviani GL, Esposito K, Morganti R, Cortelli P; Diabetic Neuropathy Study Group of the Italian Society of Diabetology. Recommendations for the use of cardiovascular tests in diagnosing diabetic autonomic neuropathy. Nutr Metab Cardiovasc Dis. 2011 Jan;21(1):69-78. doi: 10.1016/j.numecd.2010.07.005. PMID 21247746
- [Background] Lin K, Wei L, Huang Z, Zeng Q. Combination of Ewing test, heart rate variability, and heart rate turbulence analysis for early diagnosis of diabetic cardiac autonomic neuropathy. Medicine (Baltimore). 2017 Nov;96(45):e8296. doi: 10.1097/MD.0000000000008296. PMID 29137013
- [Background] Liu G, Li M, Vasanji A, Daneshgari F. Temporal diabetes and diuresis-induced alteration of nerves and vasculature of the urinary bladder in the rat. BJU Int. 2011 Jun;107(12):1988-93. doi: 10.1111/j.1464-410X.2010.09840.x. Epub 2010 Nov 18. PMID 21087392
- [Background] Beshay E, Carrier S. Oxidative stress plays a role in diabetes-induced bladder dysfunction in a rat model. Urology. 2004 Nov;64(5):1062-7. doi: 10.1016/j.urology.2004.06.021. PMID 15533519
- [Derived] Martonosi AR, Pazmany P, Kiss S, Zsakai A, Szabo L. INvesTigating the Abnormality of detrusor ConTractility by uroflowmetry in diabetic children (INTACT Trial): protocol of a prospective, observational study. BMJ Open. 2022 Nov 14;12(11):e062198. doi: 10.1136/bmjopen-2022-062198. PMID 36375985